CLINICAL TRIAL: NCT04051515
Title: Home-based vs Intradialysis Exercise Program Guided by Nursing Staff
Brief Title: Home-based vs Intradialysis Exercise Guided by Nursing Staff
Acronym: HoBIDnurse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital de Manises (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HoBIDnurse
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Exercise; Hemodialysis
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two exercise groups, intradialysis or home-based program
Who Masked: Investigator, Outcomes Assessor
Masking Description: A team of assessors, different from the researchers implementing the exercise, will record all dependent variables. A blind researcher will randomize participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradialysis exercise guided by nursing staff (Experimental): During 16 weeks subjects will exercise during the hemodialysis session, the exercise will include both aerobic and resistance training. Guidance will be provided by nursing staff
  Interventions: Other: Intradialysis exercise training
- Home-based exercise program (Active Comparator): During 16 weeks subjects will exercise on their own at home. A booklet will be provided, with a diary. Instructions to do resistance exercise with intervals of walking will be provided. Initial training will be provided by physiotherapy staff from the hospital.
  Interventions: Other: Home-based exercise training

INTERVENTIONS:
Other: Intradialysis exercise training — Combined exercise, aerobic and resistance training, implemented by nursing staff
  Arms: Intradialysis exercise guided by nursing staff
Other: Home-based exercise training — Combined exercise, aerobic and resistance training, implemented independently home
  Arms: Home-based exercise program

SUMMARY:
Participants will be randomized either to home-based exercise or to intradialysis exercise guided by nurses of the renal unit. The programs will last 16 weeks. The intradialysis exercise consists of combined aerobic and resistance training exercise. The home-based exercise consists of resistance exercise and walking.

DETAILED DESCRIPTION:
During 16 weeks one group will follow an intradialysis exercise program. The exercise program consists of strengthening exercises for lower limbs and for the upper limb free of fistula. The exercise program includes isotonic exercises for quadriceps, triceps surae, psoas, glutei, and brachial biceps; and isometric exercises for hip adductors and hamstrings. Elastic bands will be used to apply resistance. Progression will be achieved by increasing from 1 set of 10 repetitions until 3 sets of 15 repetitions. This first part of the exercise session will last no more than 30 minutes. The program will also include aerobic exercise (cycling) for up to 30 minutes. Intensity will adapted through the duration of the study so that the participant feel the exercise from hard to somewhat hard (13 to 15 at the rate of perceived exertion 6 to 20). Time and resistance will be adapted progressively. After an initial training period by a physiotherapist, the nursing staff will be responsible for monitoring and implementing the program.

The other group will follow a home-based program. A booklet with resistance exercise and recommendation of walking between exercises will be provided. An initial training phase will be applied by the physiotherapists from the rehabilitation department.

ELIGIBILITY:
Inclusion Criteria:

Patients on hemodialysis medically stable, be able to walk at least a few steps, even if you need walking aids like canes or a walker. Life expectancy greater than 6 months

Exclusion Criteria:

1. Myocardial infarction in the previous 6 weeks
2. Angina unstable on exercise or at rest
3. Brain injury derived from a cardiovascular problem. Cerebral vascular disease such as stroke in the last 6 months or with relevant sequelae in lower limb mobility presenting hemiparesia.
4. Life expectancy less than 6 months
5. Cognitive impairment
6. Language barriers
7. Illiteracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline short physical performance battery at 16 weeks | Baseline, 16 weeks
  Score achieved at the battery that includes balance tests (4 points), sit to stand to sit 5 (4 points) and and gait speed (4 points). The total score is calculated , from 1 to 12, being 12 the highest functional score
Change from baseline gait speed at 16 weeks | Baseline, 16 weeks
  Speed to cover 4 meters, in meters/second

SECONDARY OUTCOMES:
Change from baseline sit to stand 10 test at 16 weeks | Baseline, 16 weeks
  Time to perform 10 repetitions sit to stand
Change from baseline sit to stand 60 test at 16 weeks | Baseline, 16 weeks
  Sit to stand repetitions performed in 60 seconds
Change from baseline 6 minutes walk test at 16 weeks | Baseline, 16 weeks
  Number of meters walked in 6 minutes
Change from baseline handgrip strength at 16 weeks | Baseline, 16 weeks
  Bilateral handgrip strength
Change from baseline one-leg heel rise test at 16 weeks | Baseline, 16 weeks
  Number of heel rise repetitions achieved
Change from baseline one-leg standing test at 16 weeks | Baseline, 16 weeks
  Time achieved while standing on one leg
Change from baseline timed up and go test at 16 weeks | Baseline, 16 weeks
  Time to stand up, walk 3 meters, come back and sit down again
Change from baseline Physical activity level at 16 weeks | Baseline, 16 weeks
  Physical activity questionnaires
Change from baseline Health related quality of life at 16 weeks | Baseline, 16 weeks
  Medical outcomes survey Short Form 36 questionnaire to measure health-related quality of life, rated from 0 to 100, being the highest score the better the quality of life
Adherence, as number of sessions performed /number of sessions offered | 16 weeks
  Sessions performed/sessions offered

CONTACTS AND LOCATIONS:
Overall Officials: Eva Segura-Ortí, PhD, Principal Investigator — Universidad CEU Cardenal Herrera, UCH CEU
Locations (7):
- KU Leuven, Leuven, Belgium
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Spain (3):
  - Hospital de Manises, Manises, Valencia
  - Universitat de Valencia, Valencia
  - Universiat de Valéncia, Valencia
- Sweden (2):
  - Skane Univeristy Hospital, Lund
  - Karolinska Institute, Stockholm

REFERENCES:
- [Background] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637
- [Background] Segura-Orti E, Johansen KL. Exercise in end-stage renal disease. Semin Dial. 2010 Jul-Aug;23(4):422-30. doi: 10.1111/j.1525-139X.2010.00766.x. PMID 20701722
- [Background] Segura-Orti E. [Exercise in haemodyalisis patients: a literature systematic review]. Nefrologia. 2010;30(2):236-46. doi: 10.3265/Nefrologia.pre2010.Jan.10229. Epub 2010 Jan 21. Spanish. PMID 20098466
- [Background] Ortega-Perez de Villar L, Martinez-Olmos FJ, Junque-Jimenez A, Amer-Cuenca JJ, Martinez-Gramage J, Mercer T, Segura-Orti E. Test-retest reliability and minimal detectable change scores for the short physical performance battery, one-legged standing test and timed up and go test in patients undergoing hemodialysis. PLoS One. 2018 Aug 22;13(8):e0201035. doi: 10.1371/journal.pone.0201035. eCollection 2018. PMID 30133445